CLINICAL TRIAL: NCT05906316
Title: A Prospective, Multicenter, Single-arm MAC-PD Cohort: a NTM-NET and ESGMYC Collaborative Study
Acronym: MAC-PD cohort
Status: Recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-13742
Record Dates: First submitted 2023-06-07; First posted 2023-06-15 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2024-11

CONDITIONS: Mycobacterium Avium Complex Pulmonary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To gain insight in the effectiveness of, adherence and adjustments to guideline-based three-drug antimycobacterial therapy in patients with Mycobacterium avium complex pulmonary disease (MAC-PD) during the first 6 months of treatment.

DETAILED DESCRIPTION:
Mycobacterium avium complex (MAC) is the most frequent causative species that results in nontuberculous mycobacterial pulmonary disease (NTM-PD). Current treatment outcomes for MAC-PD are unsatisfactory with sputum culture conversion rates between 50-70%.The high prevalence of drug toxicity and low adherence to guideline-based treatment (GBT) are key reasons for the limited treatment success. Hence, there is an unmet need for prospective data on effectiveness of, adherence and adjustments to MAC-PD treatment regimens. By collaborating with NTM-NET and ESGMYC affiliated medical centers, we enable systematic, prospective data collection of an international MAC-PD cohort.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed MAC-PD (primary or recurrent) as per the international NTM guideline that requires three-drug antimycobacterial treatment
* Signed and dated informed consent

Exclusion Criteria:

* The participant is in poor general condition where participation in the study cannot be accepted per discretion of the Investigator
* The participant has a known or suspected, current drug or alcohol abuse, that is, in the opinion of the Investigator, sufficient to compromise the safety or cooperation of the patient
* HIV-infection;
* Cystic fibrosis;
* >1 month antibiotic treatment for current MAC infection;
* < 6 months between previous antimycobacterial NTM-PD treatment and antimycobacterial treatment for current MAC-PD
* Disseminated MAC infection;
* Active pulmonary tuberculosis, fungal or nocardial disease requiring treatment;
* Active pulmonary malignancy (primary or metastatic) or any other malignancy requiring chemotherapy or radiotherapy within 6 months before screening or anticipated during the study period;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Mycobacterium avium complex pulmonary disease that (MAC-PD) requires guideline-based three-drug antimycobacterial therapy. MAC is the most common causative species of pulmonary NTM infections.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Culture conversion rate | 6 months
  Conversion from positive cultures at baseline to negative cultures after 6 months of antimycobacterial treatment, defined by three or more negative sputum cultures sampled a month apart or one negative culture from a bronchial lavage.

SECONDARY OUTCOMES:
Change in mycobacterial load compared to baseline | 6 months
  Change in acid fast bacilli (AFB) smear determined by auramine staining
Change in mycobacterial load compared to baseline | 6 months
  Change in time-to-positivity of positive cultures
Change in symptoms compared to baseline | 6 months
  Change in symptoms as judged by the treating physician
Adverse drug reactions to antimycobacterial treatment | 6 months
  Adverse drug reactions and the (assumed) causative antimycobacterial drug
Antimycobacterial treatment adjustments | 6 months
  Any change in the antimycobacterial treatment including the reason
Other treatment adjustments | 6 months
  Changes in concomitant medication, supportive care measures or a surgical intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jakko van Ingen, MSc, PhD, Principal Investigator — Radboud University Medical Center
Locations (11):
- Oregon Science and Health University, Portland, Oregon, United States
- UZ Leuven, Leuven, Belgium
- University of Calgary, Calgary, Alberta, Canada
- University Hospital Center Zagreb, Zagreb, Croatia
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Rasmus Rude Laub, Hellerup
- University Hospital Frankfurt, Frankfurt, Germany
- Fukujuji Hospital, Tokyo, Japan
- Radboud University Medical Center, Nijmegen, Netherlands
- Seoul National University Hospital, Seoul, South Korea
- Hospital Clínic de Barcelona, Barcelona, Spain